CLINICAL TRIAL: NCT04326283
Title: A Sequential Dose-Escalation, Randomized, Active-Controlled, Multi-Center, Phase 1/2a Clinical Trial to Evaluate the Safety, Tolerability and Efficacy of SNR1611 in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Trial of Safety, Tolerability and Efficacy of Trametinib (SNR1611) in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated as it is considered that necessary data have been collected
Sponsor: Genuv Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT1SNR1611ALS1
Record Dates: First submitted 2020-03-24; First posted 2020-03-30 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Lou Gehrig's disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — trametinib; Riluzole

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned 4:1 to receive SNR1611 (0.5, 1 mg) or riluzole as an active comparator. The study will initiate with the first group of patients who will receive SNR1611 (0.5 mg, 8 patients) or riluzole (100 mg, 2 patients), while the initiation of the next dose groups will be decided by the IDMC (Independent Data Monitoring Committee) through safety assessment of the first 4-week periods of prior dose groups.
Who Masked: Outcomes Assessor
Masking Description: K-ALSFRS-R score will be measured by independent outcome assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Trametinib (0.5 mg) (Experimental): One tablet of trametinib 0.5 mg per day
  Interventions: Drug: Trametinib (0.5 mg)
- Trametinib (1 mg) (Experimental): Two tablets of trametinib 0.5 mg per day
  Interventions: Drug: Trametinib (1 mg)
- Riluzole (100 mg) (Active Comparator): One tablet of riluzole 50 mg taken twice per day
  Interventions: Drug: Riluzole (100 mg)

INTERVENTIONS:
Drug: Trametinib (0.5 mg) — 0.5 mg/day
  Other Names: Meqsel; SNR1611
  Arms: Trametinib (0.5 mg)
Drug: Trametinib (1 mg) — 1 mg/day
  Other Names: Meqsel; SNR1611
  Arms: Trametinib (1 mg)
Drug: Riluzole (100 mg) — 100 mg/day (50 mg twice)
  Other Names: Yooritek
  Arms: Riluzole (100 mg)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of trametinib (SNR1611) in the treatment of amyotrophic lateral sclerosis.

DETAILED DESCRIPTION:
Trametinib (SNR1611) is a MEK inhibitor that downregulates the MAPK/ERK pathway. In this study, the potential of MAPK/ERK pathway downregulation through trametinib (SNR1611) as a therapeutic treatment for amyotrophic lateral sclerosis (ALS) will be evaluated.

ELIGIBILITY:
Main inclusion criteria:

* Patients diagnosed as definite, probable or probable-laboratory-supported ALS according to El Escorial Criteria.
* Patients of less than 2 years after the onset of ALS.
* Patients who meet the criteria of K-ALSFRS-R score and forced vital capacity.

Main exclusion criteria:

* Patients with primary lateral sclerosis, progressive muscular atrophy or lower motor neuron disease.
* Patients who have history of ALS treatment of edaravone or stem cell therapy within 16 weeks before screening.
* Patients who have permanently ceased the administration of riluzole due to lack of tolerability and/or efficacy.
* Patients in Class II to IV according to the New York Heart Association functional classification. Patients with myocardial infarction, unstable arrhythmia, and/or significant cardiovascular disease such as unstable angina within 12 weeks before screening.
* Patients who do not meet the criteria of laboratory tests and medical/operation history.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of SNR1611: adverse events | 24-week (24-week extension and additional 48-week are optional)
  Observation of adverse events

SECONDARY OUTCOMES:
K-ALSFRS-R score | 24-week (24-week extension and additional 48-week are optional)
  Change in Korean Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (K-ALSFRS-R) score from baseline
FVC | 24-week (24-week extension and additional 48-week are optional)
  Change in Forced Vital Capacity (FVC) from baseline
CSF trough concentrations of SNR1611 | 24-week (24-week extension and additional 48-week are optional)
  Trough concentrations of SNR1611 in cerebrospinal fluid (CSF)
Plasma trough concentrations of SNR1611 | 24-week (24-week extension and additional 48-week are optional)
  Trough concentrations of SNR1611 in plasma
Milestone | Additional 48-week (optional)
  Time to event milestones

CONTACTS AND LOCATIONS:
Overall Officials: Byoung Joon Kim, Principal Investigator — Samsung Medical Center, Seoul, Republic of Korea
Locations (5):
- South Korea (5):
  - Inje University Busan Paik Hospital, Busan
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul

IPD SHARING:
Plan to Share IPD: No